CLINICAL TRIAL: NCT07370090
Title: The Effect of Self-Compassion and Self-Efficacy on Postural Awareness, Pain, and Health-Promoting Lifestyle Behaviors in Older Adults
Brief Title: Self-Compassion, Self-Efficacy, and Health Outcomes in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ACU-FTR-AOA3
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Older Adults (65 Years and Older); Health Behavior; Self-Compassion; Self-Efficacy; Pain
Keywords: Self-compassion; Self-efficacy; Older adults; Postural awareness; Health-promoting lifestyle; Pain
MeSH Terms: conditions — Health Behavior; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults: Adults aged 65 years and older who complete self-report questionnaires assessing self-compassion, self-efficacy, postural awareness, pain, quality of life, and health-promoting lifestyle behaviors.
  Interventions: Other: Questionnaire Assessment

INTERVENTIONS:
Other: Questionnaire Assessment — Participants complete validated self-report questionnaires to assess self-compassion, self-efficacy, postural awareness, pain, quality of life, and health-promoting lifestyle behaviors. No therapeutic or behavioral intervention is applied.

SUMMARY:
This cross-sectional observational study aims to examine the relationship between self-compassion, self-efficacy, postural awareness, pain, quality of life, and health-promoting lifestyle behaviors in adults aged 65 years and older. Data will be collected using validated self-report questionnaires administered online. The findings are expected to contribute to a better understanding of psychological factors associated with physical and behavioral health outcomes in older adults.

DETAILED DESCRIPTION:
Aging is associated with increased physical challenges, chronic pain, postural changes, and psychological stress. Psychological resources such as self-compassion and self-efficacy may play a protective role in maintaining both mental and physical health in older adults.

This cross-sectional observational study will recruit older adults aged 65 years and above. Participants will complete validated questionnaires assessing self-compassion, self-efficacy, postural awareness, pain, health-promoting lifestyle behaviors, and quality of life. Statistical analyses will include correlation and regression models to examine associations and predictors of pain and health-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older
* Able to read and understand Turkish
* Able to complete online questionnaires independently
* Provided informed consent

Exclusion Criteria:

* Diagnosis of severe cognitive impairment (e.g., dementia or Alzheimer's disease)
* Severe psychiatric disorders (e.g., schizophrenia or bipolar disorder)
* Inability to complete questionnaires independently
* Incomplete or inconsistent questionnaire responses

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults aged 65 years and above who are able to complete online self-report questionnaires independently.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Self-compassion level | At baseline
  Self-compassion will be assessed using the Self-Compassion Scale, a validated self-report questionnaire that evaluates individuals' compassionate attitude toward themselves across multiple dimensions.
Self-efficacy level | At baseline
  Self-efficacy will be assessed using the The Self-Efficacy Scale, which measures an individual's belief in their ability to cope with a variety of challenging demands in life.

SECONDARY OUTCOMES:
Postural awareness | At baseline
  Postural awareness will be evaluated using the Postural Awareness Scale, a self-report instrument assessing awareness of body posture and posture-related attentional regulation.
Pain severity | At baseline
  Pain severity will be assessed using the Geriatric Pain Measure, a multidimensional questionnaire designed to evaluate pain intensity and pain-related functional impact in older adults.
Health-promoting lifestyle behaviors | At baseline
  Health-promoting lifestyle behaviors will be assessed using the Health-Promoting Lifestyle Profile, which evaluates behaviors related to physical activity, nutrition, stress management, health responsibility, interpersonal relations, and self-actualization.
Quality of life score | At baseline
  Quality of life will be assessed using the WHOQOL-BREF questionnaire, which evaluates physical, psychological, social, and environmental domains of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University Kerem Aydınlar Campus, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided